CLINICAL TRIAL: NCT04693403
Title: A Multicentre, Randomized, Clinical Trial of Respiratory Support With Standard Low Flow Oxygen Therapy, Continuous Positive Airway Pressure, and High-flow Oxygen Therapy in Adults With Acute Hypoxemic Respiratory Failure in Uganda
Brief Title: The Acute Respiratory Intervention StudiEs in Africa (ARISE-AFRICA) Study
Acronym: ARISE-AFRICA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makerere University (Other)
Collaborators: THRiVE (Unknown); Paris 12 Val de Marne University (Other); Wellcome Trust (Other)
Responsible Party: Principal Investigator, College of Health Sciences, Principal Investigator, Makerere University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARISE_001
Record Dates: First submitted 2020-12-06; First posted 2021-01-05 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Acute Respiratory Failure With Hypoxia; Acute Respiratory Distress Syndrome; Acute Lung Injury
Keywords: Acute Hypoxemic Respiratory Failure; Acute Respiratory Distress Syndrome; CPAP; HFNC; Low Income Countries
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury; Respiratory Insufficiency | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: Stepped wedge cluster randomised trial (8 Clusters).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- High-flow oxygen nasal cannula (HFNC) (Experimental): In the high-flow-nasal cannula group, oxygen will be delivered through a heated humidifier and applied continuously through large-bore bi-nasal prongs, with a gas flow rate of 40-60 liters per minute and adjusted based on the clinical response.
  Interventions: Procedure: HFNC
- Continuous positive airway pressure (CPAP) (Experimental): Patients assigned to the CPAP plus oxygen group will receive periods of CPAP in addition to the standard treatment. CPAP will be started at 7.5 cm of water. The level will be decreased to 5 cm of water or increased to 10 cm of water as needed based on the clinical response and tolerance.
  Interventions: Procedure: CPAP
- Standard Low flow Oxygen Arm (Active Comparator): Patients assigned to the standard treatment group will receive oxygen delivered through a Non-rebreather face mask until endotracheal intubation, death, or fulfillment of oxygen delivery cessation criteria (an oxygen saturation by pulse oximetry (SpO2) above 92% without oxygen and a respiratory rate below 25 cycles/min).
  Interventions: Procedure: Standard Oxygen

INTERVENTIONS:
Procedure: HFNC — 40-60l/min humidified oxygen by nasal cannula
  Other Names: High-flow oxygen by nasal cannula
  Arms: High-flow oxygen nasal cannula (HFNC)
Procedure: CPAP — Oxygen therapy by boussignac Continuous positive airway pressure face mask
  Other Names: Continuous positive airway pressure
  Arms: Continuous positive airway pressure (CPAP)
Procedure: Standard Oxygen — Oxygen therapy by low flow (upto 15l/min) by Non-rebreather face mask
  Other Names: Standard Oxygen Therapy (low flow)
  Arms: Standard Low flow Oxygen Arm

SUMMARY:
The dearth of Intensive care units in low resource settings portends for poor outcomes amongst patients with acute hypoxemic respiratory failure (AHRF) . To our knowledge, the effect of CPAP and HFNC on major outcomes has not been assessed in adults with AHRF in resource-limited settings. The aim of this prospective, multicenter, randomized, controlled, trial is to determine whether High-flow oxygen through a nasal cannula (HFNC) or Continuous positive airway pressure (CPAP) system can reduce mortality among patients with acute hypoxemic respiratory failure (AHRF) in a limited resource setting as compared with standard low flow oxygen therapy?

DETAILED DESCRIPTION:
The care for the critically ill patient typically takes place in the intensive care unit (ICU). ICU care is quite expensive, even in resource rich countries. The most common reason for ICU admission globally is respiratory support for acute hypoxemic respiratory failure (AHRF). In patients with AHRF, the need for invasive mechanical ventilation is associated with high mortality, especially in low income countries (LICs), given the scarce availability of invasive mechanical ventilation. Some studies suggest that administration of ventilatory support through a mask may be effective in resource-limited settings. However, there is no clinical study data in adults to support this evidence. Human and material constraints are major barriers for the care of critically-ill patients in resource limited settings , advocating the need for a frugal approach. Furthermore, the scarcity of intensive care unit care in LICs contributes to a high mortality among acutely ill patients. The current corona virus pandemic has further highlighted the need for frugal acute care interventions in LICs.

Continuous positive airway pressure (CPAP) is a simple to use and affordable technique for noninvasive ventilatory support. High-flow oxygen through a nasal cannula (HFNC) may also offer an alternative in patients with hypoxemia. The high flow rates may also decrease physiological dead space by flushing expired carbon dioxide from the upper airway, a process that potentially explains the observed decrease in the work of breathing.

Frugal CPAP or HFNC , as compared with standard oxygen therapy, could reduce the mortality among adults presenting with AHRF in a resource-limited setting.

ELIGIBILITY:
Inclusion Criteria:

* De novo acute respiratory distress, as defined by dyspnea, use of accessory respiratory muscles, and a respiratory rate of 25 breaths per minute or more,
* Hypoxemia, as defined by a ratio of the partial pressure of arterial oxygen (PaO2) to the fraction of inspired oxygen (FiO2) of less than 300 mm Hg or a oxygen saturation by pulse oximetry SpO2/FiO2 ratio <315 will be considered for inclusion
* Informed consent obtained in accordance with local regulations;

Exclusion Criteria:

* Exacerbation of asthma, chronic obstructive pulmonary disease or another known or suspected chronic respiratory disease;
* Absolute contraindications to CPAP or HFNC
* Cardiac arrest; severe ventricular arrhythmia; shock defined by the need for vasopressors (dopamine > 5 microg/kg/min or adrenaline or noradrenaline at any dose)
* Altered consciousness (Coma Glasgow Score below 12 points);
* Do not intubate order, do not resuscitate order, or decision to limit full care taken before obtaining informed consent;
* Refusal to participate, prior enrolment in the trial, participation in another interventional study on respiratory distress;

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 705 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Mortality | 28 day
  Number of study participants deceased at day 28 of study randomisation

SECONDARY OUTCOMES:
Number of patients intubated and ventilator-free | 28 days
  Number of patients intubated and ventilator-free at 28 days from randomisation
Patient Tolerance to CPAP or HFNC | 7 days
  Patients will be assessed using the Likert scale
Organ failure free days | 7 days
  Number of days from randomisation free of organ failure
Number of patients who meet criteria for intubation at day 7 | 7 days
  Number of patients who meet criteria for intubation at day 7 of randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Kwizera, MD, Principal Investigator — Makerere University
Locations (17):
- Uganda (17):
  - Entebbe Regional Referral Hospital, Entebbe
  - St Mary's, Lacor, Gulu
  - Hoima Regional referral Hospital, Hoima
  - Jinja Regional Referral Hospital, Jinja
  - Kabale Regional Referral Hospital, Kabale
  - Mulago National Specialised Hospital, Kampala
  - Kampala hospital, Kampala
  - Kiruddu National referral Hospital, Kampala
  - Naguru Referral Hospital, Kampala
  - Nsambya Hospital, Kampala
  - Rubaga Hospital, Kampala
  - TMR International Hospital, Kampala
  - Kisoro District Hospital, Kisoro
  - Masaka regional Referral Hospital, Masaka
  - Mbale Regional referral Hospital, Mbale
  - Mbarara Regional referral Hospital, Mbarara
  - Mengo Hospital, Mengo

IPD SHARING:
Plan to Share IPD: Yes
De-identified data, upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Upon study completion, in perpetuity.
Access Criteria: By email.

REFERENCES:
- [Derived] Kwizera A, Kabatoro D, Owachi D, Kansiime J, Kateregga G, Nanyunja D, Sendagire C, Nyakato D, Olaro C, Audureau E, Mekontso Dessap A. Respiratory support with standard low-flow oxygen therapy, high-flow oxygen therapy or continuous positive airway pressure in adults with acute hypoxaemic respiratory failure in a resource-limited setting: protocol for a randomised, open-label, clinical trial - the Acute Respiratory Intervention StudiEs in Africa (ARISE-AFRICA) study. BMJ Open. 2024 Jul 1;14(6):e082223. doi: 10.1136/bmjopen-2023-082223. PMID 38951007
- See also: Related Info — https://bmjopen.bmj.com/content/14/6/e082223.info